CLINICAL TRIAL: NCT04290806
Title: Clinical Research Platform For Molecular Testing, Treatment, Quality Of Life And Outcome Of Patients With Esophageal, Gastric Or Gastroesophageal Junction Cancer Requiring Palliative Systemic Therapy
Brief Title: Registry Platform Gastric/Esophageal Cancer (SAPHIR)
Acronym: SAPHIR
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-090358
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: neoplasms; registry; health services research; epidemiology; Germany; palliative treatment; palliative care
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ESCC: 250 patients with esophageal squamous cell carcinoma
  Interventions: Other: Routine care as per site standard
- GAC: 920 patients with gastric adenocarcinoma
  Interventions: Other: Routine care as per site standard
- GEJAC: 580 patients with gastroesophageal junction adenocarcinoma
  Interventions: Other: Routine care as per site standard
- EAC: 150 patients with esophageal adenocarcinoma
  Interventions: Other: Routine care as per site standard

INTERVENTIONS:
Other: Routine care as per site standard — Physician's choice according to patient's needs. Routine care as per site standard.

SUMMARY:
The registry aims to collect and analyse information on the antineoplastic treatment of patients with metastatic esophageal, gastric or gastroesophageal junction cancer, treated in palliative intention in daily routine practice in Germany.

DETAILED DESCRIPTION:
SAPHIR is a national, observational, prospective, longitudinal, multicenter cohort study (tumor registry platform) with the purpose to record information on the antineoplastic treatment of metastatic esophageal, gastric or gastroesophageal junction Cancer in Germany. The registry will follow patients for up to two years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

Health-related quality of life (HRQoL) will be evaluated for up to two years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage IV (metastatic) ESCC, EAC, GAC or GEJAC
* Planned palliative systemic first-line therapy
* Age >= 18 years
* Signed informed consent (IC)

  * Patients answering questionnaires: IC before first therapy cycle
  * Patients not answering questionnaires: IC latest 4 weeks after start of first therapy cycle

Exclusion Criteria:

* No systemic therapy for ESCC, EAC, GAC or GEJAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic (stage IV) esophageal squamous cell carcinoma (ESCC), esophageal adenocarcinoma (EAC), gastric adenocarcinoma (GAC) or gastroesophageal junction adenocarcinoma (GEJAC), requiring palliative systemic first-line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality) | 2 years per patient
  Documentation of anamnestic data and therapy sequences

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dechow, Prof., Study Chair — Ravensburg; Florian Lordick, Prof., Study Chair — Leipzig; Sylvie Lorenzen, Prof., Study Chair — München; Karin Potthoff, Dr., Study Chair — Freiburg; Anke Reinacher-Schick, Prof., Study Chair — Bochum
Locations (1):
- Multiple sites, Gemany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No